CLINICAL TRIAL: NCT04991610
Title: Sex Determination From Scapula Using 3-D Computed Tomography in Sample of Sohag Governorate Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Daila Mohamed Khalaf, Teaching Assistant, Department of Forensic Medicine and Toxicology, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-07-15
Record Dates: First submitted 2021-07-25; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Sex Discrimination
MeSH Terms: conditions — Sexism

STUDY DESIGN:
Intervention Model Description: All measurements will be made by scanning of patients who coming to radiology department at sohag university hospital known of their birth date and sex who underwent thoracic CT scan evaluation during a pulmonary screening program . a descriptive comparative study will be conducted on total population of 100 sohag subjects (50 adult males and 50 adult females) from 25 years and above , using CT scan images to estimate the above mentioned diameters..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult male (Active Comparator): CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.
  Interventions: Radiation: computed tomography
- Adult female (Active Comparator): CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.
  Interventions: Radiation: computed tomography

INTERVENTIONS:
Radiation: computed tomography — CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.

SUMMARY:
One of the most difficult areas of forensic science is identifying individuals. Accurate sex estimation based on measurements of dimorphic dimensions in unknown human remains is a crucial first step toward making individual identification.

the most accurate approach to determine sex by bone size is based on os coxae or skull. After natural disaster their presence can never be guaranteed, therefore the development of methods of sex determination using other skeletal elements is crucial.

The scapula is a paired short bone that will be researched in this study. The decision to focus on the scapula was made in the first place because of its minor morphological alterations after growing is complete. Second, short and flat bones appear to be better maintained than lengthy bones, which are frequently fractured, scattered, and mixed together.

Scapular muscle attachments provide protection to the bone making it difficult to fracture or break .

Comparative studies on different populations have shown population-specific results in the discriminant function equations for sex estimation.

There is significant population variation due to sexual dimorphism in the growth rate and developmental process of human beings. Genetics play an important role in this variation. Nevertheless, environmental factors, nutrition, secular changes and diseases also play an important role in sexual dimorphism .

DETAILED DESCRIPTION:
One of the most difficult areas of forensic science is identifying individuals. Accurate sex estimation based on measurements of dimorphic dimensions in unknown human remains is a crucial first step toward making individual identification. the most accurate approach to determine sex by bone size is based on os coxae or skull. After natural disaster their presence can never be guaranteed, therefore the development of methods of sex determination using other skeletal elements is crucial.The scapula is a paired short bone that will be researched in this study. The decision to focus on the scapula was made in the first place because of its minor morphological alterations after growing is complete. Second, short and flat bones appear to be better maintained than lengthy bones, which are frequently fractured, scattered, and mixed together. Comparative studies on different populations have shown population-specific results in the discriminant function equations for sex estimation. There is significant population variation due to sexual dimorphism in the growth rate and developmental process of human beings. Genetics play an important role in this variation. Nevertheless, environmental factors, nutrition, secular changes and diseases also play an important role in sexual dimorphism. The first study that used the scapula in sex estimation was conducted by Dwight in 1894.

Dwight measured the height of the glenoid fossae and maximum scapular length of 123 patients (84 males and 39 females),Dwight's method showed that the scapular height had a high predictive value.

In 2010, Dabbs and Moore-Jansen applied the 23 parameter method to 803 individuals of the Hamann-Todd collection in their study and showed that the overall accuracy of this method was 95.7%.

studies reveal that the use of Computed tomography (CT) images increases accuracy and reproducibility over traditional methods in establishing a biological profile .

even though there is evidence of sexual dimorphism in the scapula according to several published studies, the validity of scapula for sex estimation has not been explored in depth in modern population where a general lack of contemporary osteometric databases noted.

in this paper , this study is presented in order to test the efficacy of scapula to serve as sex indicator for forensic purposes.

ELIGIBILITY:
Inclusion Criteria:

• persons above 25 years old

Exclusion Criteria:

* Cases below 25 years
* scapular, vertebral fractures
* growth disorders
* severe osteoporosis
* tumor
* arthritis
* previous orthopedic surgery
* infection

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — shoud be above 25 years and be healthy.
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Maximum scapular length | 12 Months
  the parameter measured The length between the highest point of superior angle and lowest point of inferior angle via software program . All CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.
Scapular breadth | 12 Months
  the parameter measured from the middle of the dorsal border of glenoid fossa to the end of spinal axis on the vertebral border. via software program All CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.
Maximum length of spine | 12 Months
  the parameter measured From the medial border of the scapula at the spinous axis to the most lateral point on the scapular spine via software program . All CT scans will be obtained from patients lying in a supine position using 120 kV tube voltage, 150 effective mA and 1 mm slice thickness parameters.

CONTACTS AND LOCATIONS:
Overall Officials: maha A Helal, professor, Study Director — faculty of medicine sohag university
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The present study aims to investigate sexual dimorphism of the scapula and establish metric standards and databases for sex estimation in a Sohag population sample
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: in july 2023
Access Criteria: Data will be gathered and analyzed using the mean, mode, and standard deviation by using SPSS program to compare mean differences between the sexes. The statistical difference will be done to compare two groups of parametric data by student - t-test .

REFERENCES:
- [Background] O'Bright L, Peckmann TR, Meek S. Is "Latin American" population-specific? Testing sex discriminant functions from the Mexican tibia on a Chilean sample. Forensic Sci Int. 2018 Jun;287:223.e1-223.e7. doi: 10.1016/j.forsciint.2018.03.046. Epub 2018 Apr 4. PMID 29692330
- [Background] Ubelaker DH, DeGaglia CM. Population variation in skeletal sexual dimorphism. Forensic Sci Int. 2017 Sep;278:407.e1-407.e7. doi: 10.1016/j.forsciint.2017.06.012. Epub 2017 Jun 19. PMID 28698063
- [Background] Papaioannou VA, Kranioti EF, Joveneaux P, Nathena D, Michalodimitrakis M. Corrigendum to "Sexual dimorphism of the scapula and the clavicle in a contemporary Greek population: Applications in forensic identification" [Forensic Sci. Int. 217 (2012) 231.e1-231.e7]. Forensic Sci Int. 2017 Jan;270:183. doi: 10.1016/j.forsciint.2016.12.012. Epub 2016 Dec 16. No abstract available. PMID 27992821